CLINICAL TRIAL: NCT02029352
Title: Topical Sinecatechins Ointment in Treatment of Primary Superficial Basal Cell Carcinoma: a Double Blind, Randomized, Placebo-controlled Trial.
Brief Title: Topical Green Tea Ointment in Treatment of Superficial Skin Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Will-Pharma (Unknown); Medigene AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL47392.068.13
Record Dates: First submitted 2013-12-18; First posted 2014-01-07 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2015-06

CONDITIONS: Carcinoma, Basal Cell
Keywords: Treatment; Sinecatechins
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — green tea extract polyphenone E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sinecatechins 10% (Experimental): Patients are instructed to apply a thin layer of the sinecatechins 10% ointment twice daily (morning and evening) in a thin layer to the tumour including 5mm of the surrounding skin. Before applying a new layer patients are advised to wipe off the remnants. Sinecatechins 10% ointment has to be applied for six weeks. Patients are advised to wash their hands after each application to prevent spreading of the ointment.
  Interventions: Drug: Sinecatechins 10%
- Placebo (Placebo Comparator): Patients are instructed to apply a thin layer of the placebo ointment twice daily (morning and evening) in a thin layer to the tumour including 5mm of the surrounding skin. Before applying a new layer patients are advised to wipe off the remnants. Sinecatechins 10% ointment has to be applied for six weeks. Patients are advised to wash their hands after each application to prevent spreading of the ointment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sinecatechins 10%
  Other Names: Veregen
  Arms: Sinecatechins 10%
Drug: Placebo — Composition, apart from the active substance, is otherwise identical to the investigational medical product.
  Arms: Placebo

SUMMARY:
Basal cell carcinoma (BCC) is the most frequently occurring nonmelanoma skin cancer in Caucasians, representing approximately 80% of cases. Incidence rates for men and women in the Netherlands are 165 and 157 per 100,000 person-years respectively and are still rising 3-10% annually. In 2009, the lifetime risk for developing a first histologically confirmed BCC for men was approximately 1 in 5 (21%) and for women it was 1 in 6 (18%).

A simplified classification of BCC includes the following three histological subtypes: nodular (40,6), superficial (30,7%) and infiltrative BCC (28,7%). Superficial BCCs (sBCCs) differ from the other subtypes as they tend to appear at a younger age, usually occur on the trunk and are often multiple. This subtype has the fastest growing incidence.

A characteristic feature of BCCs is their low risk to metastasize, though if untreated they may induce considerable functional and cosmetic morbidity as they are locally invasive. Surgery is the first treatment of choice for BCC. However due to the rising incidence and the extensive workload this entails, a non-invasive topical treatment is often chosen for sBCC as they grow down from the epidermis into the superficial dermis and therefore are easily accessible for topical treatment. Photodynamic therapy (PDT), imiquimod cream or 5-fluorouracil cream are available topical treatments for sBCC however their tumour free survival rates are not equal to the higher tumour free survival rates of surgical treatment. Next to the efficacy, the now available topical treatments are associated with local skin reactions at the treatment site, mainly erythema and erosion (imiquimod cream and 5-fluorouracil cream) or pain and burning sensation (PDT). This creates the need for additional or alternative non-invasive topical treatments.

The active constituents of green tea are promising as they are supported to have anti-BCC-carcinogenesis effects by several epidemiological, cell culture and animal studies. The so-called polyphenols known as catechins are the active constituents of green tea and the catechin epigallocatechin-3-gallate (EGCG) is the major and most active catechin. EGCG is thought to have a cytotoxic effect on skin cancer cells and has the availability of inhibition of cell growth and induction of apoptosis. It is also suggested that EGCG plays a role in inactivation of β-catenin signalling, an important component of the WNT pathway.

Sinecatechins 10% ointment (Veregen®) is a standardized extract of green tea leaves of the species Camellia sinensis, containing mainly green tea polyphenols, particularly catechins (more than 85%). The lead catechin in sinecatechins ointment is EGCG. It is approved by the US Food and Drug Administration (FDA) for genital warts in adults.

There are no clinical trials on human subjects with topical EGCG on sBCC yet. With this trial we are the first to try to validate the anti-carcinogenic potentials of topical EGCG in humans with sBCC. We assess the effectiveness of sinecatechins 10% (Veregen®) versus placebo for the topical treatment of sBCCs.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Primary histological proven superficial basal cell carcinoma ≥ 4mm and ≤ 20mm
* Comorbidities may not interfere with study treatment (evaluated by investigator)
* Capable to understand instructions

Exclusion Criteria:

* Recurrent sBCC (previous treatment)
* Breast-feeding or pregnant women
* Serious comorbidities
* Use of immunosuppressive medication during the trial period or within 30 days before enrolment
* Patients with genetic skin cancer disorders
* Tumour located in the H zone (high-risk area of face) or scalp

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-11; Primary Completion 2015-09 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with complete histological clearance | After 6 weeks treatment
  Therapeutic surgical excision of the target tumour will be performed eight weeks after start of study treatment, for histological evaluation of response.

SECONDARY OUTCOMES:
Number of applications actually done by the patient divided by the total prescribed number of applications. | Week 6
Number of local skin reactions, adverse events and serious adverse events | Up to 3 weeks
  Objective local skin signs (ie. Erythema, edema, induration, vesicles, erosion/ulceration, or other) will be assessed by the investigator at 3, 6 and 8 weeks after start of treatment.
  Subjective symptoms (ie. Pain, burning, itching, or other) will be assessed from a personal diary kept by patients once a week during treatment.
  Adverse events other than local skin reactions at the application site reported by the patient will be assessed according to the same grading.
  Other adverse events or (suspected) (unexpected) serious adverse events will be recorded by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole WJ Kelleners-Smeets, MD, PhD, Principal Investigator — Maastricht University Hospital
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Katiyar SK, Matsui MS, Elmets CA, Mukhtar H. Polyphenolic antioxidant (-)-epigallocatechin-3-gallate from green tea reduces UVB-induced inflammatory responses and infiltration of leukocytes in human skin. Photochem Photobiol. 1999 Feb;69(2):148-53. PMID 10048310
- [Background] Singh T, Katiyar SK. Green tea polyphenol, (-)-epigallocatechin-3-gallate, induces toxicity in human skin cancer cells by targeting beta-catenin signaling. Toxicol Appl Pharmacol. 2013 Dec 1;273(2):418-24. doi: 10.1016/j.taap.2013.09.021. Epub 2013 Oct 3. PMID 24096034
- [Background] Tyring SK. Effect of Sinecatechins on HPV-Activated Cell Growth and Induction of Apoptosis. J Clin Aesthet Dermatol. 2012 Feb;5(2):34-41. PMID 22468171
- [Background] Yang GY, Liao J, Kim K, Yurkow EJ, Yang CS. Inhibition of growth and induction of apoptosis in human cancer cell lines by tea polyphenols. Carcinogenesis. 1998 Apr;19(4):611-6. doi: 10.1093/carcin/19.4.611. PMID 9600345